CLINICAL TRIAL: NCT04029558
Title: Pilot Study of Nutritional Intervention, Randomized, Double Blind and Controlled Parallel Groups to Evaluate the Effect of the Consumption of the Combination of Plant Extracts (BSL_EP024) on the Immune Response in Adults
Brief Title: Effect of a Combination of Plant Extracts (BSL_EP024) on the Immune Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosearch S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C024
Record Dates: First submitted 2019-07-22; First posted 2019-07-23 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-07

CONDITIONS: Immune Response
Keywords: Immune response; Plant extracts; Dietary supplement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination of plant extracts (BSL_EP024) (Experimental): The volunteers will take two capsules daily with a combination of plant extracts (BSL_EP024)
  Interventions: Dietary Supplement: Combination of Plant Extracts (BSL_EP025)
- Placebo (Placebo Comparator): The volunteers will take two capsules daily with maltodextrin.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Combination of Plant Extracts (BSL_EP025) — Each participant will consume 2 capsules daily at lunch for 8 weeks.
  Arms: Combination of plant extracts (BSL_EP024)
Dietary Supplement: Placebo — Each participant will consume 2 capsules daily at lunch for 8 weeks.
  Arms: Placebo

SUMMARY:
The aim of the present trial is to study the effect of the combination of plant extracts (BSL_EP024) in the activation of the immune response.

DETAILED DESCRIPTION:
More than 90% of the diseases are related, directly or indirectly, with immune alterations. Traditionally, protection against infections and improvement of the immune response has been addressed by natural means through the use of plant extracts. This activity has been attributed to phenolic compounds.

The aim of the present study is to evaluate the effect of the combination of plant extracts (BSL_EP024) on immunological response parameters.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult between 18 and 55 years.
* Accept freely to participate in the study and sign the informed consent document.

Exclusion Criteria:

* Be under pharmacological treatments that may affect the immune response (anti-inflammatory drugs of chronic or frequent use, antiallergic treatments).
* Have allergy to some plant extracts
* Suffer from gastric problems or ulcers.
* Receive treatment with anticoagulant activity.
* Have a low expectation of adherence to the study protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-03 (Actual)

PRIMARY OUTCOMES:
IgM | 4 weeks
  Immunoglobulin M plasma levels
IgA | 4 weeks
  Immunoglobulin A plasma levels
IgG | 4 weeks
  Immunoglobulin G plasma levels

SECONDARY OUTCOMES:
IL-2 | 4 weeks
  Plasma levels of interleukin-2
IL-8 | 4 weeks
  Plasma levels of interleukin-8
TNF-alpha | 4 weeks
  Plasma levels of tumor necrosis factor alpha

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Quesada, MD, PhD, Study Chair — Medical specialist in Endocrinology, Hospital San Cecilio de Granada
Locations (1):
- Biosearch Life, Granada, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No